CLINICAL TRIAL: NCT01574976
Title: Effect of Feedback and Practice on Probabilistic Decision Making in Attention Deficit and Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Yehuda Pollak, clinical neuropsychologist, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 37/12
Record Dates: First submitted 2012-04-01; First posted 2012-04-10 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: ADHD
Keywords: ADHD; probabilistic; choice; feedback; practice
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- control, no feeback (Active Comparator): subjects without ADHD, probabilistic choices without feedback
  Interventions: Behavioral: probabilistic choice
- control, feedback (Active Comparator): subjects without ADHD, probabilistic choices with feedback
  Interventions: Behavioral: probabilistic choice
- ADHD, no feedback (Experimental): subjects with ADHD, probabilistic choices without feedback
  Interventions: Behavioral: probabilistic choice
- adhd, feedback (Experimental): subjects with ADHD, probabilistic choices with feedback
  Interventions: Behavioral: probabilistic choice

INTERVENTIONS:
Behavioral: probabilistic choice — subjects should choose between low-certain outcome and high-uncertain outcome

SUMMARY:
The purpose of this study is to determine how feedback and practice affect decision making in adolescents with attention deficit and hyperactivity disorder.

Participants will have to choose between low and certain outcome and a higher but uncertain outcome, with or without serial feedback after each trial. Participants will perform the task twice to examine practice effects.

ELIGIBILITY:
Inclusion Criteria:

* ADHD

Exclusion Criteria:

* Current major depression,
* Psychosis,
* Autism,
* Tourette syndrome

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
probabilistic choice | 1 year
  The number of risky outcomes a subject chose on a probabilistic choice paradigm

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Pollak, PhD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel, Israel